CLINICAL TRIAL: NCT02984163
Title: The Alberta Cancer Exercise "ACE" Program for Cancer Survivors: Supporting Community-based Exercise Participation for Health Promotion and Secondary Cancer Prevention
Brief Title: Alberta Cancer Exercise Hybrid Effectiveness-Implementation Study
Acronym: ACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other); Alberta Health services (Other); Cross Cancer Institute (Other); Tom Baker Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-16-0905
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Neoplasms
Keywords: cancer; exercise
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Intervention (Experimental): Participant exercise sessions will be conducted in groups of 10-15 under the direct supervision of the community-based exercise specialist. Sessions will be twice a week for 12-weeks. Participants will have the option to continue with the exercise program after the 12-weeks on a fee-for-service basis.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise sessions will include a combination of aerobic, resistance, balance, and flexibility exercises delivered in a circuit-type class setting or group personal training format.
  Other Names: Physical Activity

SUMMARY:
The primary purpose of this proposed 5-year hybrid effectiveness and implementation study is to evaluate the relative benefit from, and implementation of an Alberta wide clinic-to-community-based cancer and exercise model of care - the Alberta Cancer Exercise (ACE) Program. The investigators hypothesize that the strategy will improve the physical well-being and QoL of survivors (on and off cancer treatment) while preventing the development of secondary cancers.

DETAILED DESCRIPTION:
A total of 2500 adult cancer survivors will be enrolled in the 5-year study. The investigators will build capacity by expanding ACE training and programming to sites beyond the large urban centers. The investigators plan for implementation in 7 Alberta YMCAs and/or City Recreation facilities within 3 years, as well as to formally establish partnerships within AHS to build further capacity across the province within existing AHS programming (e.g., CancerControl Rehab Services, Alberta Healthy Living Program and Primary Care Network). Virtual and supported home-based options will be available as an alternative.

Eligible and consenting participants will be screened for exercise safety, and following fitness testing will be triaged to appropriate exercise programming in their home or community. The exercise intervention will take place at the survivor's home, YMCAs and municipal fitness centres across the province. The supported home-based and community-based exercise program will be administered by exercise specialists who have undergone the ACE Cancer and Exercise: Training for Fitness Professionals course. Survivors will take part in a combination of aerobic, resistance, balance, and flexibility exercises delivered in a circuit-type class setting or group personal training format, twice weekly for an 8-to-12-week period.

Effectiveness outcomes include physical fitness, physical activity, quality of life, and healthcare utilization. These outcomes are known factors associated with the secondary prevention of cancer. The RE-AIM framework will be used to evaluate program reach, effectiveness, adoption, implementation and maintenance. The Alberta Quality Matrix for Health will serve as a framework to inform program sustainability beyond the funding period. Through this research, the investigators will better understand the effectiveness of the ACE program, and evaluate processes to support future implementation and sustainability.

ELIGIBILITY:
Inclusion Criteria:

1. have a diagnosis of cancer;
2. be over the age of 18 years;
3. be able to participate in low-intensity levels of activity at minimum;
4. be pretreatment, or receiving active cancer treatment (i.e., surgery, systemic therapy and radiation therapy), or have received cancer treatment within the past 3 years; or have ongoing significant cancer or treatment-related impairments (requiring supportive exercise intervention);
5. be able to provide informed written consent in English.

Exclusion criteria:

1) Inability or deemed unsafe to participate in physical activity program

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2570 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Minutes Per Week | Baseline to One-year
  Change in number of participants meeting Guidelines for Physical Activity of 150 minutes per week of moderate intensity exercise

SECONDARY OUTCOMES:
Aerobic Endurance | Baseline to One-year
  Change in 6 minute walk test distance (metres)
Quality of Life Cancer Specific | Baseline to One year
  Change in Functional Assessment of Cancer Therapy General Scale
General Health-related Quality of Life | Baseline to One-year
  Change in Rand Short Form (SF)-36
Fatigue | Baseline to One-year
  FACT-Fatigue subscale
Upper extremity grip strength | Baseline to One-year
  Change in hand-grip dynamometry (kg)
Functional performance test | Baseline to One-year
  Change in sit-to-stand (number in 30 seconds)
Upper extremity flexibility | Baseline to One-year
  Change in active shoulder flexion range of motion (degrees)
Lower extremity flexibility | Baseline to One-year
  Change in sit-and-reach test (cm)
Balance | Baseline to One-year
  Change in one legged stance test (seconds)
Cost-effectiveness evaluation | Baseline to One-year
  EQ-5D questionnaire
Exercise adherence | Baseline to 12-weeks
  Adherence to exercise programming (attendance at sessions)
Body Composition | Baseline to One-year
  Change in BMI
Waist and hip measurements | Baseline to One-year
  Change in waist and hip circumference (cm) and change in waist-to-hip ratio
Program implementation and evaluation | Baseline to One-year
  RE-AIM: program reach, effectiveness, adoption, implementation and maintenance
Adverse events | Baseline to One-year
  Adverse event rates

OTHER OUTCOMES:
Home-based programming stepping test | Baseline to One-year
  2-minute stepping test
1RM or 8RM strength (optional) | Baseline to One-year
  Change in bench press, vertical row and leg press strength (kg)
Muscular endurance test (optional) | Baseline to One-year
  Change in number of push-ups
Core endurance test (optional) | Baseline to One-year
  Change in plank test (seconds held)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L McNeely, PT, PhD, Principal Investigator — University of Alberta; Nicole Culos-Reed, PhD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary/ Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta & Cross Cancer Institute, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Undecided
No plan in place at this point in time.

REFERENCES:
- [Derived] McNeely ML, Sellar C, Williamson T, Shea-Budgell M, Joy AA, Lau HY, Easaw JC, Murtha AD, Vallance J, Courneya K, Mackey JR, Parliament M, Culos-Reed N. Community-based exercise for health promotion and secondary cancer prevention in Canada: protocol for a hybrid effectiveness-implementation study. BMJ Open. 2019 Sep 13;9(9):e029975. doi: 10.1136/bmjopen-2019-029975. PMID 31519676